CLINICAL TRIAL: NCT02141659
Title: A Phase 1, Open-label, Multicenter Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of TAK-385 Alone in Hormone Treatment- naïve Japanese Patients With Non-metastatic Prostate Cancer
Brief Title: A Study of TAK-385 in Hormone Treatment-naïve Participants With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-385/TB-AK160108; U1111-1156-6034 (Registry Identifier: WHO)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Hormone Treatment-naïve Participants With Prostate Cancer
MeSH Terms: interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg (Experimental): TAK-385 320 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 80 mg maintenance dose, tablet, orally, once daily through Days 2 to 28.
  Interventions: Drug: TAK-385
- Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg (Experimental): TAK-385 320 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 120 mg maintenance dose, tablet, orally, once daily through Days 2 to 28.
  Interventions: Drug: TAK-385
- Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg (Experimental): TAK-385 320 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 160 mg maintenance dose, tablet, orally, once daily through Days 2 to 28.
  Interventions: Drug: TAK-385
- Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg (Experimental): TAK-385 360 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 120 mg maintenance dose, tablet, orally, once daily through Days 2 to 28.
  Interventions: Drug: TAK-385
- Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg (Experimental): TAK-385 320 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 80 mg maintenance dose, tablet, orally, once daily through Days 2 to 672.
  Interventions: Drug: TAK-385
- Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg (Experimental): TAK-385 320 mg loading dose, tablet, orally, once on Day 1, followed by TAK-385 120 mg maintenance dose, tablet, orally, once daily through Days 2 to 672.
  Interventions: Drug: TAK-385

INTERVENTIONS:
Drug: TAK-385 — TAK-385 Tablets.

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of TAK-385 in hormone treatment-naïve participants with non-metastatic prostate cancer.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the tolerability and safety of TAK-385 in hormone treatment-naive participants with non-metastatic prostate cancer. This study consists of two parts: Part A, multiple dose-rising (MRD) phase and Part B, an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participants judged by the investigator to have the capacity to understand the study and follow the study rules.
2. Participants whose written consent (signature or printed name and personal seal on informed consent form) can be obtained before any study procedures are performed.
3. Japanese male participants 20 or more years of age at the time of informed consent.
4. Participants who, if they have a female partner who could become pregnant, agree to practice appropriate means of contraception from the time of informed consent throughout the entire study treatment period and for 4 months after the last dose of study drug.
5. Participants in stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks (28 days) prior to study treatment initiation.
6. Participants with histologically or cytologically confirmed prostate cancer.
7. Participants whose clinical diagnosis is T1-4 N0 M0, or Tx N0 M0 for participants who have undergone radical prostatectomy.
8. Participants who are considered eligible for hormone therapy for prostate cancer.
9. Participants who have not received hormone therapy (example, gonadotropin-releasing hormone [GnRH] agonist, GnRH antagonist, steroidal antiandrogen, non-steroidal androgen) for prostate cancer.
10. Participants who have not undergone surgical castration.
11. Participants with serum testosterone at screening greater than (>) 150 nanogram per deciliter (ng/dL).
12. Participants meeting either of the following criteria for prostate-specific antigen (PSA) at screening. Untreated prostate cancer: PSA at screening > 4.0 nanogram per milliliter (ng/mL) Treated* prostate cancer: PSA at screening > 0.2 ng/mL.

    * Participants who have undergone prostatectomy or either or both of high intensity focused ultrasound therapy or radiotherapy (excluding 125I-brachytherapy) prior to the start of this study.
13. Eastern Cooperative Oncology Group (ECOG) Performance Status [17] of 0 or 1.
14. Body mass index (BMI) at screening greater than or equal to (>=) 18.0 kilogram per square meter (kg/m^2).

Exclusion Criteria:

1. Participants exhibiting symptoms judged related to prostate cancer by the investigator (example, bone pain, pelvic pain, ureteral obstruction) who urgently require hormone therapy such as GnRH agonist, GnRH antagonist, or CAB/MAB therapy, chemotherapy, or radiotherapy.
2. Participants who have received 5-alpha reductase inhibitors (except for participants who have been treated for male-pattern alopecias).
3. Participants who have received chemotherapy for prostate cancer (including estramustine).
4. Participants who have received 125I-brachytherapy.
5. Participants who received radiotherapy (except for 125I-brachytherapy) within 16 weeks (112 days) before study treatment initiation.
6. Participants who underwent prostatectomy within 16 weeks (112 days before study treatment initiation.
7. Treatment with any investigational compound within the 4 weeks (28 days) prior to the first dose of study drug or ongoing participation in another experimental trial related to the treatment of prostate cancer.
8. Diagnosis or treatment for another systemic malignancy within 2 years before study treatment initiation, or who had received a diagnosis of another malignancy before that and have evidence of residual disease. Participants with non-melanoma skin cancer or carcinoma in situ who have undergone complete resection will not be excluded from the study.
9. Participants taking drugs with moderate to strong cytochrome P450 3A4 (CYP3A4) inhibitory or inducing effects, or any medications, supplements, or food products with P-glycoprotein (P-gp) inhibitory effects, in the 2 weeks (14 days) prior to study treatment initiation.
10. Participants who have received TAK-385 in a past clinical study.
11. Participants for whom it would be difficult to collect blood from a peripheral vein.
12. Participants with uncontrolled and clinically significant nervous, circulatory, pulmonary, hepatic, renal, metabolic, gastrointestinal, urogenital, or endocrine disorders, or other abnormalities (except for the targeted disease) that could affect study participation or the study results. Also, participants meeting any of criteria a through c below.

    A. Participants with uncontrolled diabetes (Hemoglobin A1c [HbA1C] > 8 percent [%] at screening). However, participants whose HbA1c is brought under control with diabetes medications may be rescreened.

    B. Participants with uncontrolled hypertension (systolic blood pressure > 150 millimeter of mercury (mmHg) and diastolic blood pressure > 90 mmHg at 2 separate measurements taken no more than 60 minutes apart at screening). Participants whose blood pressure is brought under control by antihypertensive medication may be rescreened.

    C. Participants with myocardial infarction, unstable symptomatic ischemic heart disease, arrhythmias of common terminology criteria for adverse events (CTCAE) Grade > 2, thromboembolism (deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or other heart diseases (example, pericardial effusion, restrictive cardiomyopathy). However, chronic stable atrial fibrillation controlled by stable anticoagulant therapy will be allowed.
13. Participants with bilateral hydronephrosis or bladder neck outlet obstruction.
14. Known hypersensitivity to TAK-385, TAK-385 excipients, or gonadotropin-releasing hormone (GnRH) antagonists.
15. Participants with a past history of gastrointestinal tract treatments (including gastrectomy) or gastrointestinal disease that could affect the drug absorption or tolerability (malabsorption, esophageal reflux, peptic ulcer, erosive esophagitis).
16. Participants positive for hepatitis B surface antigens (HBsAg), hepatitis C antibodies (HCV), human immunodeficiency virus (HIV) antibodies, or serologic test for syphilis, or with life-threatening disease other than cancer, at screening.
17. Clinically relevant electrocardiogram (ECG) abnormalities, or the following ECG abnormalities, at screening.

    * Q-wave infarction, unless identified 6 or more months prior to TAK-385 treatment initiation.
    * QTcF interval > 450 millisecond (msec) (when calculating the QTc interval, Fridericia's equation [QT/RR0.33] will be used).
18. Participants with congenital QT prolongation.
19. Current use of Class 1A or Class 3 antiarrhythmic medications.
20. New York Heart Association Class III or IV heart failure.
21. Participants with clinical laboratory abnormalities suggesting clinically relevant underlying disease, or with any of the following abnormal results, at screening.

    * Serum creatinine >= 2.0 mg/dL.
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >= 1.5*upper limit of normal (ULN) for the study site.
    * Total bilirubin >= 2*ULN for the study site.
    * Neutrophil count less than (<) 1,500 per cubic millimeter (/mm^3), platelet count < 100,000 per microliter (/mcL), hemoglobin < 10.0 g/dL.
    * Results of heart-related tests (creatine kinase MB [CK-MB] and cardiac troponin T) exceeding the study sites reference value.
22. Participants found to have clinical problems on the basis of examination findings, ECG findings, or chest X-ray findings at screening.
23. Participants considered unlikely by investigators to be able to follow the study protocol or considered ineligible for the study by investigators for other reasons.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Japan (6):
  - Sakura-shi, Chiba
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Chiyoda-ku, Tokyo

REFERENCES:
- [Derived] Suzuki H, Uemura H, Mizokami A, Hayashi N, Miyoshi Y, Nagamori S, Enomoto Y, Akaza H, Asato T, Kitagawa T, Suzuki K. Phase I trial of TAK-385 in hormone treatment-naive Japanese patients with nonmetastatic prostate cancer. Cancer Med. 2019 Oct;8(13):5891-5902. doi: 10.1002/cam4.2442. Epub 2019 Aug 19. PMID 31429205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Japan from 01 May 2014 to 20 April 2017.
Pre-assignment Details: Japanese participants with hormone treatment-naive prostate cancer were enrolled in this study to receive TAK-385 loading dose (320 or 360 milligram [mg]) and maintenance dose (80, 120 or 160 mg) in two parts: Part A, dose-escalation phase, cohorts 1-4 and Part B, dose-expansion phase, cohorts 1-2.
Period: Overall Study
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Started | 3 | 4 | 3 | 3 | 15 | 15
Completed | 3 | 3 | 3 | 3 | 13 | 13
Not Completed | 0 | 1 | 0 | 0 | 2 | 2
Not completed — Major Protocol Deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pretreatment Event/ Adverse Event | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 15 | 15 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  years | 73.3 (5.51) | 72.0 (5.60) | 75.0 (6.08) | 71.7 (3.51) | 74.5 (4.84) | 74.4 (5.53) | 74.0 (5.00)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 3 | 4 | 3 | 3 | 15 | 15 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  participants
    Japan | 3 | 4 | 3 | 3 | 15 | 15 | 43
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  centimeter (cm) | 166.0 (5.57) | 167.0 (3.92) | 162.3 (3.06) | 160.3 (4.16) | 163.4 (3.94) | 164.7 (5.27) | 164.1 (4.57)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  kilogram (kg) | 63.27 (8.361) | 64.40 (9.542) | 57.97 (2.857) | 56.80 (1.992) | 64.43 (7.891) | 59.34 (5.440) | 61.59 (7.017)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The safety analysis set included all participants who received at least 1 dose of study drug.
  kilogram per square meter (kg/m^2) | 22.90 (2.100) | 23.03 (2.841) | 22.00 (1.400) | 22.17 (1.498) | 24.17 (3.109) | 21.93 (2.475) | 22.90 (2.694)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as treatment-related adverse events (AEs) that occurred within the first 28 days of treatment as per common terminology criteria for adverse events (CTCAE) version 4.03: any grade 3 or higher toxicity; QT/Fridericia corrected QT (QTcF) greater than (>) 500 millisecond (msec) after treatment initiation; QT/QTcF interval prolongation >60 msec postdose.
Time Frame: From treatment initiation until Day 28
Population: The DLT analysis set included all participants enrolled in cohort A that meeting the following; who had taken at least 80 percent (%) of the doses of TAK-385 (23 doses) during the DLT evaluation period and for whom the DLT evaluation period observations had been completed or who had experienced DLTs during the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants Reporting One or More Treatment-emergent Adverse Event (TEAE)
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 68)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 4 | 3 | 3
Participants | 3 | 2 | 3 | 2

3. Primary Outcome: Part A: Number of Participants With Grade 2 or Higher Laboratory Test Abnormalities
Description: Laboratory test abnormalities were graded using the CTCAE. The grades were: Grade 2- (moderate) minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activity of daily living (ADL); Grade 3- (severe) medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care ADL. Data has been presented for any Grade 2 or higher event in the laboratory test abnormalities.
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 68)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 4 | 3 | 3
Participants
  Grade 2: White Blood Cell Low | 1 | 0 | 0 | 1
  Grade 2: Neutrophil Count Low | 0 | 0 | 0 | 1
  Grade 2: Lymphocyte Count Low | 1 | 1 | 0 | 0
  Grade 2: Potassium Low | 0 | 0 | 1 | 0

4. Primary Outcome: Part A: Number of Participants With Markedly Abnormal Values of Vital Signs Parameters
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 68)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 4 | 3 | 3
Participants
  Body Temperature <35.6 degree Celsius | 1 | 1 | 0 | 0
  Systolic BP >180 millimeter of Mercury (mmHg) | 1 | 0 | 0 | 0
  Diastolic BP <50 mmHg | 1 | 0 | 0 | 0
  Pulse <50 beats per minute (bpm) | 1 | 1 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Markedly Abnormal Values of Electrocardiogram (ECG) Parameters
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 68)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 4 | 3 | 3
Participants
  Heart Rate <50 bpm | 1 | 2 | 0 | 0
  QT Interval >=460 millisecond (msec) | 1 | 2 | 0 | 1

6. Primary Outcome: Part B: Number of Participants Reporting One or More TEAE
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 712)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

7. Primary Outcome: Part B: Number of Participants With Grade 2 or Higher Laboratory Test Abnormalities
Description: Laboratory test abnormalities were graded using the CTCAE. The grades were: Grade 2- (moderate) minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL; Grade 3- (severe) medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care ADL. Data has been presented for any Grade 2 or higher event in the laboratory test abnormalities. Here aspartate aminotransferase (AST) (glutamic-oxaloacetic transaminase [GOT]) High, creatine kinase (CK) (creatine phosphokinase [CPK]) High, prothrombin time (PT)-international normalized ratio (INR) High.
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 712)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
Participants
  Grade 2: White Blood Cell Low | 1 | 3
  Grade 3: White Blood Cell Low | 1 | 0
  Grade 3: Hemoglobin Low | 1 | 0
  Grade 2: Neutrophil Count Low | 2 | 2
  Grade 2: Lymphocyte Count Low | 1 | 1
  Grade 3: Lymphocyte Count Low | 1 | 0
  Grade 2: Glucose High | 2 | 2
  Grade 3: Bilirubin Total High | 0 | 1
  Grade 2: AST (GOT) High | 1 | 0
  Grade 2: Gamma-glutamyl Transferase (GGT) High | 2 | 0
  Grade 2: CK (CPK) High | 2 | 1
  Grade 2: Potassium Low | 1 | 1
  Grade 2: Corrected Calcium Low | 1 | 0
  Grade 2: PT- INR High | 0 | 1
  Grade 2: Triglycerides High | 1 | 1
  Grade 3: Triglycerides High | 0 | 1

8. Primary Outcome: Part B: Number of Participants With Markedly Abnormal Values of Vital Signs Parameters
Description: Here "BP" is blood pressure.
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 712)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
Participants
  Body Temperature <35.6 degree Celsius | 7 | 4
  Systolic BP >180 mmHg | 1 | 0
  Diastolic BP >110 mmHg | 1 | 0
  Diastolic BP <50 mmHg | 0 | 1
  Pulse <50 bpm | 2 | 1

9. Primary Outcome: Part B: Number of Participants With Markedly Abnormal Values of ECG Parameters
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 712)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
Participants
  Heart Rate <50 bpm | 4 | 2
  QT Interval >=460 msec | 5 | 4
  QTcF Interval >=500 msec | 2 | 5

10. Secondary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration for Unchanged TAK-385 on Day 1, 14 and 28
Time Frame: Days 1, 14 and 28 pre-dose and at multiple time points (up to 12 hours for Days 1 and 14; up to 72 hours for Day 28) post-dose
Population: The pharmacokinetic (PK) evaluable population included participants who received at least 1 dose of study drug, without major protocol deviations, and met the minimum protocol prescription. The PK analysis population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
nanogram per milliliter (ng/mL)
  Day 1 | 191.7 (94.405) | 198.0 (62.386) | 250.0 (207.56) | 254.0 (330.58)
  Day 14 | 23.53 (1.4189) | 94.40 (115.08) | 216.1 (151.78) | 65.57 (40.840)
  Day 28: number analyzed (Participants) | 3 | 3 | 2 | 3
  Day 28 | 38.10 (21.743) | 34.43 (24.962) | 94.70 (114.98) | 25.56 (16.275)

11. Secondary Outcome: Part A: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to (Tau) Over the Dosing Interval for Unchanged TAK-385 on Day 1, 14 and 28
Time Frame: as for outcome 10
Population: The PK evaluable population included participants who received at least 1 dose of study drug, without major protocol deviations, and met the minimum protocol prescription. The PK analysis population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliter (h*ng/mL)
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
hour*nanogram per milliter (h*ng/mL)
  Day 1 | 679.7 (96.340) | 933.0 (604.30) | 761.7 (249.78) | 663.3 (501.85)
  Day 14 | 199.0 (49.487) | 363.8 (291.00) | 741.7 (385.96) | 379.0 (199.65)
  Day 28: number analyzed (Participants) | 3 | 3 | 2 | 3
  Day 28 | 239.0 (75.020) | 323.4 (230.40) | 469.0 (458.21) | 227.5 (138.37)

12. Secondary Outcome: Part A: Serum Testosterone Concentrations for TAK-385
Time Frame: Up to Day 35
Population: The full analysis set included all participants who received at least 1 dose of study drug. The full analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg
Number analyzed (Participants) | 3 | 4 | 3 | 3
ng/mL
  Baseline | 5.440 (1.6829) | 6.505 (2.6175) | 6.317 (1.7503) | 7.853 (1.1885)
  Day 2: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 2 | 0.603 (0.1457) | 0.977 (0.5288) | 0.777 (0.2485) | 1.477 (1.3540)
  Day 3: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 3 | 0.350 (0.0917) | 0.460 (0.1852) | 0.483 (0.1762) | 0.623 (0.3232)
  Day 7 | 0.283 (0.0764) | 0.380 (0.2177) | 0.377 (0.1332) | 0.337 (0.0416)
  Day 14: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 14 | 0.140 (0.0173) | 0.213 (0.1102) | 0.213 (0.1012) | 0.203 (0.0379)
  Day 21: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 21 | 0.143 (0.0635) | 0.220 (0.1044) | 0.207 (0.0635) | 0.207 (0.0666)
  Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 28 | 0.137 (0.0577) | 0.200 (0.0700) | 0.190 (0.0693) | 0.243 (0.0802)
  Day 31: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 31 | 0.137 (0.0416) | 0.217 (0.1002) | 0.170 (0.0436) | 0.210 (0.0854)
  Day 35: number analyzed (Participants) | 3 | 3 | 3 | 3
  Day 35 | 0.130 (0.0436) | 0.290 (0.2433) | 0.153 (0.0321) | 0.167 (0.0473)

13. Secondary Outcome: Part B: Percent Change From Baseline in PSA Levels on Week 13 Day 1 Last Observation Carried Forward (LOCF)
Time Frame: Baseline, and Week 13 Day 1 (LOCF; up to Week 13 Day 1)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
percent change | -89.77 (13.886) | -93.91 (5.161)

14. Secondary Outcome: Part B: Plasma Concentration of Unchanged TAK-385
Time Frame: Up to Week 49 Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 14
ng/mL
  Week 1 Day 1 | 0.000 (0.0000) | 0.000 (0.0000)
  Week 1 Day 1: 2 hours postdose: number analyzed (Participants) | 14 | 12
  Week 1 Day 1: 2 hours postdose | 72.89 (123.81) | 88.58 (124.65)
  Week 1 Day 2 | 6.406 (6.0223) | 9.854 (7.4824)
  Week 1 Day 4 | 4.683 (2.7897) | 7.565 (5.0412)
  Week 2 Day 1: number analyzed (Participants) | 15 | 12
  Week 2 Day 1 | 3.972 (1.7426) | 8.146 (5.3370)
  Week 3 Day 1: number analyzed (Participants) | 15 | 13
  Week 3 Day 1 | 4.123 (2.2959) | 8.618 (6.8455)
  Week 5 Day 1: number analyzed (Participants) | 14 | 14
  Week 5 Day 1 | 4.122 (1.8301) | 9.105 (6.6634)
  Week 5 Day 1: 2 hours postdose: number analyzed (Participants) | 14 | 14
  Week 5 Day 1: 2 hours postdose | 20.90 (19.603) | 30.82 (35.770)
  Week 9 Day 1: number analyzed (Participants) | 14 | 14
  Week 9 Day 1 | 4.076 (2.1577) | 9.496 (6.6435)
  Week 13 Day 1: number analyzed (Participants) | 14 | 14
  Week 13 Day 1 | 4.239 (2.2374) | 9.820 (7.2860)
  Week 17 Day 1: number analyzed (Participants) | 14 | 14
  Week 17 Day 1 | 4.759 (2.9601) | 9.269 (6.2961)
  Week 21 Day 1: number analyzed (Participants) | 13 | 12
  Week 21 Day 1 | 4.254 (2.0265) | 11.08 (10.873)
  Week 25 Day 1: number analyzed (Participants) | 13 | 12
  Week 25 Day 1 | 5.592 (3.2911) | 11.95 (11.792)
  Week 37 Day 1: number analyzed (Participants) | 13 | 11
  Week 37 Day 1 | 4.924 (3.7682) | 11.32 (10.759)
  Week 49 Day 1: number analyzed (Participants) | 13 | 11
  Week 49 Day 1 | 4.683 (3.1686) | 10.08 (8.1482)

15. Secondary Outcome: Part B: Serum Testosterone Concentrations for TAK-385
Time Frame: Up to Week 97 Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
Number analyzed (Participants) | 15 | 15
ng/mL
  Baseline | 6.367 (1.9930) | 7.243 (2.2424)
  Week 1 Day 2 | 0.975 (0.5247) | 0.867 (0.5835)
  Week 1 Day 4 | 0.384 (0.0968) | 0.463 (0.2313)
  Week 2 Day 1 | 0.285 (0.0741) | 0.318 (0.1165)
  Week 3 Day 1 | 0.207 (0.0580) | 0.235 (0.0925)
  Week 5 Day 1 | 0.213 (0.0701) | 0.190 (0.0670)
  Week 9 Day 1 | 0.195 (0.0554) | 0.191 (0.0818)
  Week 13 Day 1: number analyzed (Participants) | 14 | 15
  Week 13 Day 1 | 0.209 (0.0746) | 0.181 (0.0631)
  Week 17 Day 1: number analyzed (Participants) | 14 | 15
  Week 17 Day 1 | 0.217 (0.0757) | 0.175 (0.0548)
  Week 21 Day 1: number analyzed (Participants) | 13 | 14
  Week 21 Day 1 | 0.222 (0.0844) | 0.179 (0.0794)
  Week 25 Day 1: number analyzed (Participants) | 13 | 14
  Week 25 Day 1 | 0.218 (0.0816) | 0.202 (0.1069)
  Week 37 Day 1: number analyzed (Participants) | 13 | 13
  Week 37 Day 1 | 0.229 (0.1046) | 0.208 (0.1177)
  Week 49 Day 1: number analyzed (Participants) | 13 | 13
  Week 49 Day 1 | 0.228 (0.0922) | 0.196 (0.0849)
  Week 61 Day 1: number analyzed (Participants) | 11 | 9
  Week 61 Day 1 | 0.204 (0.0823) | 0.212 (0.1111)
  Week 73 Day 1: number analyzed (Participants) | 11 | 9
  Week 73 Day 1 | 0.218 (0.0974) | 0.203 (0.1206)
  Week 85 Day 1: number analyzed (Participants) | 10 | 8
  Week 85 Day 1 | 0.253 (0.0878) | 0.259 (0.1358)
  Week 97 Day 1: number analyzed (Participants) | 10 | 8
  Week 97 Day 1 | 0.283 (0.1364) | 0.311 (0.1792)

ADVERSE EVENTS:
Time Frame: From treatment initiation until 40 days after last dose of study drug (Day 68 for Part A and Day 712 for Part B)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/3 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/3 | 3/15 | 3/15
Other Adverse Events (participants affected / at risk) | 3/3 | 2/4 | 3/3 | 2/3 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg (N=3) | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg (N=4) | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg (N=3) | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg (N=3) | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg (N=15) | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg (N=15)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Device loosening (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Cohort 1: TAK-385 320 mg + TAK-385 80 mg (N=3) | Part A Cohort 2: TAK-385 320 mg + TAK-385 120 mg (N=4) | Part A Cohort 3: TAK-385 320 mg + TAK-385 160 mg (N=3) | Part A Cohort 4: TAK-385 360 mg + TAK-385 120 mg (N=3) | Part B Cohort 1: TAK-385 320 mg + TAK-385 80 mg (N=15) | Part B Cohort 2: TAK-385 320 mg + TAK-385 120 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 2 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 2 | 0 | 0 | 2 | 6 | 9
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinea manuum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 5
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hangover (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 5
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Bone density decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Occult blood (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Listless (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scrotal mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02141659/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT02141659/SAP_001.pdf